CLINICAL TRIAL: NCT06456294
Title: Evaluation of a Medication Health Center to Promote Opioid Safety
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1840701
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Overdose
Keywords: naloxone; opioids; safety
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MHC Early Outreach Intervention (Experimental): Early implementation of a MHC outreach intervention program. Clinics in the early outreach intervention arm will be assigned to the MHC Direct patient outreach, where MHC staff will encourage patients to schedule an appointment with the MHC and primary care (PC) staff will be educated to encourage MHC visits.
  Interventions: Behavioral: MHC Outreach Intervention
- MHC Delayed Outreach Intervention (No Intervention): Clinics in the usual care/delayed intervention arm will deliver usual care through the health plan, pharmacy and clinicians. As part of usual care, patients at these clinics can access naloxone through physician prescription or standing orders.

INTERVENTIONS:
Behavioral: MHC Outreach Intervention — Adult PC clinics are randomized to receive the MHC Outreach Intervention early (n=7 clinics) vs. delayed (n=7 clinics). In early intervention clinics, patients prescribed chronic opioid therapy, on a chronic opioid registry, and receiving their medication from the intervention clinic are sent emails and letters inviting them to schedule an MHC appointment. Clinical staff at the early intervention clinic are educated to encourage attendance. During MHC visits, MHC staff assess patients prescribed Chronic Opioid Therapy (COT), educate them about overdose, prescribe naloxone, and order guideline-concordant opioid monitoring.
  Arms: MHC Early Outreach Intervention

SUMMARY:
This study will assess the impact of an opioid safety clinic intervention for patients prescribed chronic opioid therapy. Outcomes are visits to the clinic, naloxone dispensings, Prescription Drug Monitoring reviews, and Urine Drug Screens conducted

DETAILED DESCRIPTION:
Given ongoing concerns about the risk of opioid overdose among people taking chronic opioid therapy for pain, Kaiser Permanente Colorado (KPCO) sought to develop a standardized approach to promote opioid safety. Operational stakeholders adapted an existing Opioid Safety Clinic model, tailored it for KPCO's context, and implemented it in three geographically dispersed KPCO clinics with leadership support. The approach was a multidisciplinary "Medication Health Center" to assess patients, educate them about overdose risk, provide naloxone, and ensure adherence to standard monitoring. Operations and the research team then collaborated to assess the effectiveness of the program to inform decisions to scale the program to other regions.

ELIGIBILITY:
Evaluation population:

1. Eligible Clinics
2. Patients prescribed Chronic Opioid Therapy

Eligibility Criteria for Clinics:

1. Clinic leadership willing to be randomized to order of implementation
2. Not a pilot location

Eligibility for an MHC visit included the following:

1. Patients in the KPCO chronic opioid registry
2. No Primary Care Physician (PCP) or MHC visit in the past 6 months
3. Not managed by the Integrated Pain Service, a specialty pain service that takes care of the highest risk and most complex pain patients

Patients enter the chronic opioid registry if they fulfill any of the following criteria:

* 2 opioid fills in the last 90 days; fills should be separated by 27 days, or
* 1 opioid fill with pill number ≥100 pills in the last 90 days, or
* 1 long-acting/extended-release opioid fill in the last 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-12-03 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a Medication Health Center visit | Outcomes are assessed in a two-month post-intervention period.
  Medication Health Center (MHC) Visits will be assessed using data from the electronic medical record.

SECONDARY OUTCOMES:
Number of participants with a Naloxone dispensing | Outcomes are assessed in a two-month post-intervention period.
  Naloxone dispensings are assessed using data from the electronic medical record
Number of participants with a Prescription Drug Monitoring Program (PDMP) review | Outcomes are assessed in a two-month post-intervention period.
  Prescription Drug Monitoring Program (PDMP) reviews are assessed using data from the electronic medical record
Number of participants with a Urine Drug Screens completed | Outcomes are assessed in a two-month post-intervention period.
  Urine Drug Screens Completed are assessed using data from the electronic medical record

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators interested in using the data from this study must submit a written request. Requests must address regulatory and compliance requirements for data usage. Investigators must outline the necessary resources required to support their data request, including personnel and infrastructure. The original study team will evaluate each request based on scientific merit, ethical considerations, and alignment with the original study's objectives.
  Deidentified electronic health record (EHR) data will be shared with investigators upon approval of written request. Investigators are responsible for obtaining necessary approvals and adhering to relevant laws and regulations and will be required to sign a Data Use Agreement (DUA) outlining the terms and conditions of data usage. The data sharing period is limited to three years following the publication of the primary study.
Time Frame: 3 years after following publication